CLINICAL TRIAL: NCT03708783
Title: Study on Short and Long-term Outcome of Laparoscopic Spleen-Preserving No. 10 Lymph Node Dissection for Advanced Middle or Upper Third Gastric Cancer
Brief Title: Laparoscopic Spleen-Preserving No. 10 Lymph Node Dissection for AGC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xiangqian Su, Chief of GI surgery IV, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFH2018-2-2153
Record Dates: First submitted 2018-10-08; First posted 2018-10-17 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Gastric Cancer; Gastrectomy; Laparoscopic Surgery; Lymphadenectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with locally advanced upper and middle third gastric cancer will receive laparoscopic total gastrectomy with D2 lymphadenectomy including No. 10 lymph node dissection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No. 10 Lymph Node Dissection group (Experimental): Patients with locally advanced upper or middle third gastric cancer will receive laparoscopic total gastrectomy and D2 lymphadenectomy with spleen-preserving No.10 lymph node dissections
  Interventions: Procedure: laparoscopic Spleen-Preserving No. 10 Lymph Node Dissection

INTERVENTIONS:
Procedure: laparoscopic Spleen-Preserving No. 10 Lymph Node Dissection — For patients with locally advanced upper or middle third gastric cancer, laparoscopic total gastrectomy with D2 lymphadenectomy including spleen-preserving No. 10 lymph node dissection is performed.

SUMMARY:
The purpose of this study is to explore the safety and feasibility of laparoscopic spleen-preserving No. 10 lymph node dissection for patients with advanced middle or upper third gastric cancer.

DETAILED DESCRIPTION:
Radical resection is the primary treatment for patients with advanced middle or upper third gastric cancer. And D2 lymphadenectomy, including No. 10 lymph node dissection, should be performed according to the Japanese treatment guidelines for gastric cancer. Because of the complexity of the anatomy around the spleen, spleen-preserving No. 10 lymph node dissection is difficult. Although Professor Huang from Fujian Medical University Union Hospital has proposed the "Huang's three-step maneuver" to dissect No. 10 lymph node with preserved spleen laparoscopically, such method is far from popularized, especially in North China. In addition, the safety, feasibility and oncological efficacy of this method was not confirmed in such area, either.

In this study, a prospective, single center, single-arm, non-inferiority clinical trial will be conducted to evaluate the short and long-term outcome of the laparoscopic spleen-preserving No. 10 lymph node dissection for patients with locally advanced middle or upper third gastric cancer in Beijing.

ELIGIBILITY:
Inclusion Criteria:

* Patients age older than 18 years (including 18 years old);
* The primary lesion is located in the upper or middle third of the stomach, including Siewert II type and Siewert III type adenocarcinoma of the esophagogastric junction;
* Pathologically confirmed primary gastric adenocarcinoma by endoscopic biopsy (including papillary, tubular, mucinous, signet ring cell and poorly differentiated adenocarcinoma);
* Preoperative cancer stage cT2-4aN0-3M0 (according to AJCC-7th TNM staging);
* The Eastern Cooperative Oncology Group performance status of 0 or 1;
* The American Society of Anesthesiology classes of I, II or III;
* Signed Informed consent.

Exclusion Criteria:

* Pregnant or lactating women;
* Suffering from severe mental disorder;
* Previous gastrectomy, including endoscopic submucosal dissection and endoscopic mucosal resection;
* Integrated or enlarged lymph node with maximum diameter larger than 3 cm according to preoperative imaging, including significantly enlarged or bulky No. 10 lymph nodes;
* Siewert I type adenocarcinoma of the esophagogastric junction;
* Other malignant diseases (within 5 years);
* Other illnesses needed operation concurrently;
* Complications (bleeding, perforation or obstruction) required emergency surgery due to primary gastric malignancy;
* Pulmonary function tests FEV1 less than 50% of predicted value;
* Patient suffered from bleeding tendency disease such as hemophilia or took anti-coagulant medication due to deep vein thrombosis.
* Patients with obvious tumor infiltration in the spleen and splenic vessels which require splenectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of postoperative complications within 30 days | 30 days

SECONDARY OUTCOMES:
3-year disease free survival | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No